CLINICAL TRIAL: NCT00631384
Title: Experimental Design of Couple Counseling and Testing in Antenatal Clinics in Dar es Salaam, Tanzania
Acronym: CVCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: H.32.02.05.29
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: HIV Infections
Keywords: Voluntary Counseling and Testing; HIV; HIV seronegativity
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Women to be asked to bring husbands for couple VCT
  Interventions: Behavioral: Couples VCT
- 2 (Active Comparator): Women to receive individual VCT
  Interventions: Behavioral: Individual VCT

INTERVENTIONS:
Behavioral: Couples VCT — Offer women coming to antenatal clinics to have their husbands come with them for couples VCT
  Arms: 1
Behavioral: Individual VCT — Women to receive individual VCT
  Arms: 2

SUMMARY:
The objective of this research is to evaluate the effectiveness of couples Voluntary Counseling and Testing for HIV (CVCT) compared to individual VCT (IVCT) in preventing MTCT, and in increasing preventive behaviors and minimizing spousal abuse among HIV positive women. We hypothesize that offering CVCT will not decrease uptake of VCT among women. This research will be carried out in 3 antenatal clinics in Dar es Salaam, Tanzania.

ELIGIBILITY:
Inclusion Criteria:

* Up to 6 months of pregnancy
* Currently married or in cohabiting union for 2+ years and co-resident with husband

Exclusion Criteria:

* In polygamous marriage
* 7 or more months pregnant

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1521 (Actual)
Dates: Start 2003-03; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
HIV Testing and receiving results | within one month of initial visit to ANC

SECONDARY OUTCOMES:
use of nevirapine | 3 months after testing
use of protection at time of sexual intercourse | 3 months after HIV test
domestic violence | 3 months after HIV test

CONTACTS AND LOCATIONS:
Locations (1):
- Muhimbili University College of Health Sciences, Dar es Salaam, Tanzania